CLINICAL TRIAL: NCT01643798
Title: Role of the Supraspinal Opioidergic Circuit in Prefrontal TMS-Induced Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1F30DA033748 (NIH); 1F30DA033748-01 (NIH)
Record Dates: First submitted 2012-06-22; First posted 2012-07-18 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Participants received intravenous saline immediately prior to sham and real rTMS of the left dorsolateral prefrontal cortex. The parameters of the stimulation paradigm are as follows: 10 Hz, 5 seconds on, 10 seconds off, 20 minutes, 4000 pulses).
  Interventions: Procedure: Sham rTMS; Procedure: Real rTMS
- Naloxone (Active Comparator): Participants received intravenous naloxone (0.1mg/kg) immediately prior to sham and real rTMS of the left dorsolateral prefrontal cortex. The parameters of the stimulation paradigm are as follows: 10 Hz, 5 seconds on, 10 seconds off, 20 minutes, 4000 pulses).
  Interventions: Procedure: Sham rTMS; Procedure: Real rTMS

INTERVENTIONS:
Procedure: Sham rTMS — The eSham system was implemented in conjunction with a specialized Neuronetics sham TMS coil. This coil has a metal plate hidden inside of it that blocks the magnetic field from affecting the brain. Scalp electrodes were used to mimic the feel of real rTMS. This approach has been validated in previous studies.
  Other Names: Neuronetics Model 2100 Therapy System
Procedure: Real rTMS — An iron-core, solid-state figure-of-8 coil was used to stimulate the dorsolateral prefrontal cortex. The site of stimulation was estimated using the Beam F3 method based on the 10-20 EEG system.
  Other Names: Neuronetics Model 2100 Therapy System

SUMMARY:
Studies have shown that transcranial magnetic stimulation (TMS), a non-invasive form of brain stimulation, can reduce pain in the laboratory and in the clinic. The purpose of this study is to investigate how TMS relieves pain and affects pain circuitry in the brain. One of the primary study hypotheses is that opioid blockade will significantly reduce the pain relief produced by left prefrontal cortex TMS.

DETAILED DESCRIPTION:
Non-invasive forms of brain stimulation such as transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS) are currently being investigated as alternative or adjunctive therapies for pain. Clinical interest in these techniques continues to grow because of rising opiate abuse and inadequate pain management strategies. Despite this enthusiasm, studies on the efficacy of repetitive TMS (rTMS) for pain have produced mixed results. Some of the most promising and informative research has focused on rTMS for perioperative pain. In two different postoperative studies, a single session of left dorsolateral prefrontal cortex (DLPFC) rTMS after gastric bypass surgery reduced morphine self-administration by 40% when compared to sham stimulation. These data are particularly fascinating given the role of the DLPFC in top-down pain processing.

Centered at the juncture of Brodmann Areas (BAs) 9 and 46, the DLPFC remains a popular therapeutic target for rTMS given its accessible location and presumed role in high-order cognition and emotional valence. Animal and human studies suggest that cingulofrontal regions like DLPFC may modulate pain perception via recruitment of opioidergic midbrain and brainstem structures like the periaqueductal gray (PAG) and the rostroventromedial medulla (RVM), respectively. These data outline the functional circuitry that might be involved in the analgesic effects of DLPFC rTMS.

While many studies aim to evaluate the clinical efficacy of DLPFC rTMS for pain management, few have examined how it affects pain processing. Imaging the cerebral signature of pain before and after left DLPFC rTMS might reveal information about pain circuitry and help to elucidate the mechanism by which prefrontal rTMS may produce analgesia. Previous studies suggest that opioid blockade abolishes left but not right DLPFC rTMS-induced analgesia. In this study, our a priori hypothesis was that left DLPFC rTMS would attenuate blood oxygenation-level dependent (BOLD) signal response to painful stimuli in pain processing regions. More specifically, we anticipated that midbrain and medulla BOLD signal changes induced by left DLPFC rTMS would be abolished by pretreatment with the μ-opioid antagonist naloxone.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* no history of depression or pain
* no metal in body
* no medications that lower seizure threshold

Exclusion Criteria:

* history of depression or pain
* history of seizures or epilepsy
* metal implants in body
* medications that lower seizure threshold
* psychiatric medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Taylor, Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective participants were interviewed over the phone prior to being invited to a screening visit in the Brain Stimulation Laboratory at MUSC. Risks and benefits were explained and consent was obtained. All participants were tested for opiate use and females were tested for pregnancy. Recruitment began in 2011 and ended in early 2012.
Pre-assignment Details: Healthy volunteers were randomized to receive I.V. saline or naloxone immediately prior to sham and real rTMS on the same experimental visit. One week later, each participant received the novel pretreatment but the same stimulation paradigm. One participant dropped out after her first experimental visit. These data were not included.
Groups:
- Saline and Stimulation, Then Naloxone and Stimulation: Participants received an intravenous infusion of 10ml sterile saline immediately prior to sham and real rTMS of the left dorsolateral prefrontal cortex. One week later, participants received an intravenous infusion of 0.1 mg/kg Naloxone immediately prior to sham and real rTMS of the left dorsolateral prefrontal cortex
- Naloxone and Stimulation, Then Saline and Stimulation: Participants received an intravenous infusion of 0.1mg/kg Naloxone immediately prior to sham and real rTMS of the left dorsolateral prefrontal cortex. One week later, participants received an intravenous infusion of 10ml sterile saline immediately prior to sham and real rTMS of the left dorsolateral prefrontal cortex
Period: Pretreatment 1 and Stimulation
Arm/Group | Saline and Stimulation, Then Naloxone and Stimulation | Naloxone and Stimulation, Then Saline and Stimulation
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Pretreatment 2 and Stimulation
Arm/Group | Saline and Stimulation, Then Naloxone and Stimulation | Naloxone and Stimulation, Then Saline and Stimulation
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pretreatment & Stimulation: Outside of the 3T magnetic resonance imaging (MRI) scanner, participants underwent resting motor threshold assessment, left dorsolateral prefrontal cortex localization and preliminary pain testing. Next, participants were placed in the scanner for baseline pain testing. After baseline testing, participants were asked to rate the pain that they had experienced. Participants were subsequently removed from the scanner and randomized to receive approximately 10 ml intravenous naloxone (0.1mg/kg) or saline immediately prior to 20 minutes of sham left DLFPC rTMS. Following sham rTMS, participants returned to the scanner for the same block testing performed at baseline. After rating their pain, participants were removed from the scanner for 20 minutes of real left DLPFC rTMS. Participants then returned to the scanner for the final block test.
Arm/Group | Pretreatment & Stimulation
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating
Description: There are two experimental visits separated by one week. During each experiment, pain ratings will be measured every 30 minutes. "Preliminary testing" will be done 30 minutes into the experiment. The purpose of preliminary testing is to select the temperature that will be used to induce pain throughout the experiment. "Baseline testing" will be done 60 minutes into the experiment. "After sham rTMS" will be done 90 minutes into the experiment. "After real rTMS" will be done 120 minutes into the study. The pain scale used in a Visual Analog Scale (VAS). There was an 11-point rating system where "0" represented no pain and "10" represented unbearable pain.
Time Frame: Baseline (60 minutes into experiment), Post-Sham (90 minutes), Post-Real (120 minutes)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Sham rTMS With Saline; Real rTMS With Saline; Sham rTMS With Naloxone; Real rTMS With Naloxone: Participants first underwent baseline pain testing in the scanner. At the conclusion of baseline testing, participants were asked to rate the pain that they had experienced. Participants were subsequently removed from the scanner and randomized to receive 10 ml intravenous (I.V.) naloxone (0.1 mg/kg) or saline immediately before 20 min of sham left DLFPC rTMS. Following sham rTMS, participants returned to the scanner for the same block testing performed at baseline. After rating their pain, participants were removed from the scanner for 20min of real left DLPFC rTMS. Participants then returned to the scanner for the final block test. The I.V. pretreatment was randomized such that participants received saline on one visit and naloxone on the other visit.
Arm/Group | Sham rTMS With Saline | Real rTMS With Saline | Sham rTMS With Naloxone | Real rTMS With Naloxone
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale | 7.36 (0.24) | 5.61 (0.26) | 7.54 (0.15) | 6.75 (0.21)
Statistical Analysis 1: Comparison: Sham rTMS With Saline vs Real rTMS With Saline; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sham rTMS With Naloxone vs Real rTMS With Naloxone; Test type: Superiority or Other; p = 0.04, ANOVA

2. Primary Outcome: Change in BOLD Signal in Pain Processing Regions During Pain, Including Supraspinal Opioidergic Structures
Description: There are two experimental visits separated by one week. During each experiment, blood oxygen level dependent (BOLD) signal will be measured at baseline (60 minutes into the experiment), post-sham rTMS (90 minutes into the experiment) and post-real (120 minutes into the experiment).
Time Frame: Baseline (60 minutes into experiment), Post-Sham (90 minutes), Post-Real (120 minutes)
Measure: Mean (Standard Error); unit: mean percentage of BOLD signal change
Groups:
- Sham rTMS With Saline; Real rTMS With Saline; Sham rTMS With Naloxone; Real rTMS With Naloxone: Participants first underwent baseline pain testing in the scanner. At the conclusion of baseline testing, participants were asked to rate the pain that they had experienced. Participants were subsequently removed from the scanner and randomized to receive 10 ml intravenous (I.V.) naloxone (0.1 mg/kg) or saline immediately before 20 min of sham left DLFPC rTMS. Following sham rTMS, participants returned to the scanner for the same block testing performed at baseline. After rating their pain, participants were removed from the scanner for 20min of real left DLPFC rTMS. Participants then returned to the scanner for the final block test. The I.V. pretreatment was randomized such that participants received saline on one visit and naloxone on the other visit. Whole-brain and anatomical region of interest analysis were performed. The numbers below represent midbrain percent signal change.
Arm/Group | Sham rTMS With Saline | Real rTMS With Saline | Sham rTMS With Naloxone | Real rTMS With Naloxone
Number analyzed (Participants) | 14 | 14 | 14 | 14
mean percentage of BOLD signal change | 0.15 (0.03) | 0.00 (0.04) | 0.10 (0.03) | 0.13 (0.05)
Statistical Analysis 1: Comparison: Sham rTMS With Saline vs Real rTMS With Saline; Test type: Superiority or Other; p = .0003, ANOVA
Statistical Analysis 2: Comparison: Sham rTMS With Naloxone vs Real rTMS With Naloxone; Test type: Superiority or Other; p = 0.794, ANOVA

ADVERSE EVENTS:
Arm/Group | Pretreatment & Stimulation
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes